CLINICAL TRIAL: NCT05885516
Title: Double vs Single Intrauterine Insemination in Male Factor Infertility - a Multicenter Randomized Trial
Brief Title: Double vs Single Intrauterine Insemination in Male Factor Infertility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Merve Dizdar, Principal Investigator, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/384
Record Dates: First submitted 2023-05-01; First posted 2023-06-02 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Male Factor Infertility

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single intrauterine insemination group (Placebo Comparator): When the leading follicle is greater than 17 mm following ovulation induction with follicle stimulating hormone (FSH) daily injections, ovulation trigger injection will be given to the participant. 36 hours after ovulation trigger injection single intrauterine insemination with partner's sperm collected on the same day will be done.
  Interventions: Procedure: intrauterine insemination
- Double intrauterine insemination group (Experimental): When the leading follicle is greater than 17 mm following ovulation induction with follicle stimulating hormone (FSH) daily injections, ovulation trigger injection will be given to the participant. 24 and 48 hours after ovulation trigger injection intrauterine insemination will be done twice with partner's sperm collected on the specified days.
  Interventions: Procedure: intrauterine insemination

INTERVENTIONS:
Procedure: intrauterine insemination — Giving washed sperm concentrate into uterine cavity via a soft catheter

SUMMARY:
The aim of the study is to compare the pregnancy outcomes of single vs double intrauterine insemination (IUI) in couples with male factor infertility.

DETAILED DESCRIPTION:
The principle behind double intrauterine insemination in male factor infertility couples is to create a longer time frame for fertilization and to increase motile sperm number in female genital tract in order to increase pregnancy rates. There's a clinical equipoise on the benefits of performing double IUI in couples following ovarian hyperstimulation with daily follicle stimulating hormone injections in male factor subfertility. As it is stated in Cochrane database, there's a need for adequately powered, randomized, high-quality studies on this subject.

In this study, as a result of a-priori power analysis 132 participants in each study arm is planned to be recruited in the study. Male factor infertility included in the study is defined as total motile sperm count (TPMSC) less than 10 million. TPMSC less than 1 million, female age greater than 40, uterine anomaly, no patent tubes shown in hysterosalpingography, history of ovarian surgery and known endometriosis will be excluded. Couples with two basal semen analysis with TPMSC between 1-10 million will be randomized to single or double IUI procedure. To accomplish this in approximately 1 year period, the study is planned as a multi-center study.

The objective of the study is to compare the pregnancy outcomes of single and double intrauterine insemination groups, following ovarian hyperstimulation in couples with male factor subfertility.

ELIGIBILITY:
Inclusion Criteria:

* Couples trying to conceive for at least 6 months despite of regular sexual intercourse
* Female partner between 18-40 years old
* Male partner sperm analysis total motile sperm count between 1-10 million in at least 2 sperm analysis on different days.

Exclusion Criteria:

* No patent fallopian tubes shown in hystero-salpingography
* Female partner with a uterine anomaly
* History of a previous ovarian surgery
* Known or suspected endometriosis in female partner
* Body-mass index (BMI) > 40 kg/m2

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is not based on self-representation of gender identity. Participants should have a uterus with at least one patent fallopian tube and an internal os to achieve intrauterine insemination.
Enrollment: 264 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-11-22 (Estimated); Study Completion 2024-12-22 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical pregnancy | Within 4-6 weeks after insemination
  Pregnancy with fetal cardiac activity diagnosed by transvaginal ultrasonography

SECONDARY OUTCOMES:
Rate of biochemical, ectopic pregnancies and rate of miscarriages | Within 3 months after insemination
  Pregnancy outcomes including biochemical, ectopic pregnancies and miscarriages diagnosed by transvaginal ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rakic L, Kostova E, Cohlen BJ, Cantineau AE. Double versus single intrauterine insemination (IUI) in stimulated cycles for subfertile couples. Cochrane Database Syst Rev. 2021 Jul 14;7(7):CD003854. doi: 10.1002/14651858.CD003854.pub2. PMID 34260059
- [Background] Bagis T, Haydardedeoglu B, Kilicdag EB, Cok T, Simsek E, Parlakgumus AH. Single versus double intrauterine insemination in multi-follicular ovarian hyperstimulation cycles: a randomized trial. Hum Reprod. 2010 Jul;25(7):1684-90. doi: 10.1093/humrep/deq112. Epub 2010 May 10. PMID 20457669